CLINICAL TRIAL: NCT01651208
Title: Improving Adherence to Post PCI Antiplatelet Therapy in Minority Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Humana Inc. (Industry)
Responsible Party: Principal Investigator, Ana M. Palacio, Associate Professor of Clinical Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1RC1MD004327 (NIH)
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary stents; Medication adherence; Antiplatelet medications; Motivational Interviewing
MeSH Terms: conditions — Coronary Artery Disease; Medication Adherence | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational interviewing (MINT) (Experimental): The MINT intervention will consist of 4 to 7 telephone encounters between a nurse trained in Motivational interviewing and a minority subject who recently received a coronary stent. All subjects in the MINT arm will be contacted every 3 months to complete 4 encounters. MINT is a well-known, scientifically tested behavioral counseling strategy developed as an amalgamation of principles drawn from several theoretical paradigms, the most important of which are Self-Determination Theory, Patient-Centeredness, Self-Efficacy theory, and the Stages of Change model.
  Interventions: Behavioral: Motivational Interviewing (MINT)
- Mailed DVD (Active Comparator): A DVD that re-enforces an adequate behavior regarding adherence to anti-platelet will be compared to a MINT intervention. The DVD will also address many questions and concerns patients have after stent placement. The intervention is based on role theory and the effects of vicarious learning via electronic media with respect to Cardiovascular behaviors.
  Interventions: Behavioral: Mailed DVD

INTERVENTIONS:
Behavioral: Motivational Interviewing (MINT) — We will hire a Latino and an AA nurse to deliver the interventions and will match their race/ethnicity with that of the subject. Past experience suggests that at 4-7 calls per subjects each lasting about 30-45 minutes, a nurse can carry a caseload of about 125-150 subject (we propose 125 per nurse) Each telephone encounter will have a patient centered approach having the following basic structure and goals:
  a)Establishing a connection and reinforcing autonomy b)Empathizing with ambivalence and rolling with resistance.c)Coach the subject towards expressions of commitment.
  Arms: Motivational interviewing (MINT)
Behavioral: Mailed DVD — The DVD will have a documentary format that will engage subjects as the portrayed real patients relate their struggles and successes, that will entertain and ultimately motivate subjects to succeed in a similar way as the role models in the video. That personal connection will activate patients to address their own adherence issues and will show real life ways to deal with the health behaviors recommended post PCIS. Key concepts regarding adherence to medications and other behaviors will be imbedded in the story telling. The DVD will also feature a humanistic perspective of a cardiologist talking about his concerns for his patients that do not adhere to the antiplatelet therapy, the difficulties that his patients face, and the merit of the success stories he witnesses.
  Arms: Mailed DVD

SUMMARY:
The purpose of this study is to evaluate if the use of a phone based motivational interviewing among minority populations who received a coronary stent can improve adherence to antiplatelet agents from approximately 51% to 66% (15 percentage point increase) at 12 months post stent placement when compared to a mailed educational DVD.

DETAILED DESCRIPTION:
Other aims are: 1) Improve the self reported adherence of antiplatelet medications 2) Identify specific barriers for the use of post PCI anti-platelet therapy among minority populations enrolled in Humana by administering a short survey at the baseline recruitment call and at the 12 month follow up call, 3) identify predictors of never filling an anti-platelet therapy prescription post PCIS.

Inclusion criteria:

We will include black or Hispanic patients having coronary stenting using the following codes for bare metal or drug eluting stents: ICD-9 procedure codes (36.06) or (36.07), MS-DRG codes 247-249 or CPT codes 92980, 92981, C1984 G0290, G0291. The identification period will last approximately 10 months.

Primary Outcome: Medication Possession ratio as a dichotomous variable (appropriate/not appropriate adherence) and as a continuous variable

Secondary outcomes:

Self reported adherence by 4- item Morisky Medication Adherence Scale (MMAS-4) Barriers to appropriate adherence Predictors of adherence

ELIGIBILITY:
Inclusion Criteria:

* We will identify prospectively all subjects who undergo coronary stenting using the following codes for bare metal or drug eluting stents: ICD-9 procedure codes (36.06) or (36.07), MS-DRG codes 247-249 or CPT codes 92980, 92981, C1984 G0290, G0291
* We will select subjects identified as Black or Hispanics by a validated algorithm that uses the Medicare race code, geocoding techniques and the Spanish Surname list.

Exclusion Criteria:

1. Lack of medical files to document stent placement.
2. Not receiving informed consent.
3. Subjects with contraindications for antiplatelet therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Palacio, MD, MPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Background] Palacio AM, Tamariz LJ, Uribe C, Li H, Salkeld EJ, Hazel-Fernandez L, Carrasquillo O. Can claims-based data be used to recruit black and Hispanic subjects into clinical trials? Health Serv Res. 2012 Apr;47(2):770-82. doi: 10.1111/j.1475-6773.2011.01316.x. Epub 2011 Aug 30. PMID 22091834

RESULTS

PARTICIPANT FLOW:
Groups:
- Motivational Interviewing (MINT): The MINT intervention consists of quarterly telephone encounters between a nurse trained in Motivational interviewing and a minority subject who recently received a coronary stent. Each call would last approximately 30 minutes. .MINT is a well-known, scientifically tested behavioral counseling strategy developed as an amalgamation of principles drawn from several theoretical paradigms, the most important of which are Self-Determination Theory, Patient-Centeredness, Self-Efficacy theory, and the Stages of Change model.
Period: Overall Study
Arm/Group | Motivational Interviewing (MINT) | Mailed DVD
Started | 227 | 225
Completed | 213 (14 patients had no pharmacy claims data to analyze primary outcome) | 209 (16 subjects had no pharmacy claims data to analyze primary outcome)
Not Completed | 14 | 16
Not completed — Lost to Follow-up | 14 | 16

BASELINE CHARACTERISTICS:
Groups:
- Motivational Interviewing (MINT): The MINT intervention will consist of quarterly telephone encounters between a nurse trained in Motivational interviewing and a minority subject who recently received a coronary stent. .MINT is a well-known, scientifically tested behavioral counseling strategy developed as an amalgamation of principles drawn from several theoretical paradigms, the most important of which are Self-Determination Theory, Patient-Contentedness, Self-Efficacy theory, and the Stages of Change model.
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing (MINT) | Mailed DVD | Total
Number analyzed (Participants) | 227 | 225 | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.11 (8.65) | 69.94 (9.01) | 69.52 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 89 | 190
  Male | 126 | 136 | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 101 | 100 | 201
  Not Hispanic or Latino | 126 | 125 | 251
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 126 | 125 | 251
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 101 | 100 | 201
Educational level [Number; unit: participants] — Achieved high school education or higher
  participants
    High School or Higher | 51 | 49 | 100
    Less than High School | 176 | 176 | 352

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Appropriate Adherence/ Medication Possession Ratio (MPR)
Description: Medication Possession ratio (MPR) is a continuous multiple interval measure of medication availability. This is a validated method of estimating medication adherence . The medication possession ratio is defined as the sum of the days' supply of medication divided by the number of days between the first fill and the last refill plus the days' supply of the last refill.We will use the previously validated cutpoint of MPR>=.80 to define the binary outcome of Appropriate Adherence
Time Frame: 12 months after receiving coronary stent
Measure: Number; unit: participants
Arm/Group | Motivational Interviewing (MINT) | Mailed DVD
Number analyzed (Participants) | 227 | 225
participants | 137 | 105
Statistical Analysis 1: Comparison: Motivational Interviewing (MINT) vs Mailed DVD; We hypothesized that in the MINT group, at least 70% of subjects will reach an MPR of 0.80 while in the DVD group, the proportion will remain at or below 55%. Our sample size estimates showed that, using a conservative 2-sided test at the 5% Alpha level and a 90% power, we will be able to detect a significant 15% difference (70% - 55%) with a sample of 217 in each study group; Test type: Superiority or Other; p < 0.01, Chi-squared

2. Secondary Outcome: 4-Item Morisky Medication Adherence Scale (MMAS-4)
Description: The Morisky 4-Item Medication Adherence Scale (MMAS-4) is a self-reported measure of medication-taking behavior. Available in 33 languages, it addresses barriers to medication-taking. Each question can be answer as Yes or No for a range of 0-4 points.
Time Frame: At 12 month post stent placement
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Motivational Interviewing (MINT): The MINT intervention will consist of 4 to 7 telephone encounters between a nurse trained in Motivational interviewing and a minority subject who recently received a coronary stent. All subjects in the MINT arm will be contacted every 3 months to complete 4 encounters.MINT is a well-known, scientifically tested behavioral counseling strategy developed as an amalgamation of principles drawn from several theoretical paradigms, the most important of which are Self-Determination Theory, Patient-Centeredness, Self-Efficacy theory, and the Stages of Change model.
  Motivational Interviewing (MINT): Each telephone encounter will have a patient centered approach having the following basic structure
Arm/Group | Motivational Interviewing (MINT) | Mailed DVD
Number analyzed (Participants) | 227 | 225
Score on a Scale | 3.82 (.45) | 3.60 (.69)
Statistical Analysis 1: Comparison: Motivational Interviewing (MINT) vs Mailed DVD; The null hypothesis is that the mean MMAS-4 score is similar in both intervention arms; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 0.29

ADVERSE EVENTS:
Arm/Group | Motivational Interviewing (MINT) | Mailed DVD
Serious Adverse Events (participants affected / at risk) | 0/227 | 0/225
Other Adverse Events (participants affected / at risk) | 0/227 | 0/225

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No